CLINICAL TRIAL: NCT00533273
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Efficacy of AA4500 in the Treatment of Subjects With Advanced Dupuytren's Disease Followed by an Open-Label Extension Phase
Brief Title: Non-US Study of AA4500 (XIAFLEX™, Proposed Name) in the Treatment of Advanced Dupuytren's Disease
Acronym: CORD-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUX CC 859
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Results first posted 2010-10-22 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Advanced Dupuytren's Disease
MeSH Terms: interventions — Microbial Collagenase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AA4500 0.58 mg (Experimental)
  Interventions: Biological: collagenase clostridium histolyticum
- Placebo (Placebo Comparator)
  Interventions: Biological: collagenase clostridium histolyticum

INTERVENTIONS:
Biological: collagenase clostridium histolyticum — Subjects could have received up to three injections of AA4500 0.58 mg/placebo into the cord of the affected hand in the double-blind phase. In the open-label extension phase, subjects could have received up to five additional injections of AA4500, with each injection separated by at least 30 days. Individual joints could have received up to a maximum of three AA4500 injections.
  Other Names: XIAFLEX®; AA4500

SUMMARY:
This 12-month study had two phases: a 90-day double-blind, randomized, placebo-controlled phase and a nine-month open-label extension phase. Before treatment, eligible subjects were stratified by the primary joint type (30 metacarpophalangeal [MP] joints and 30 proximal interphalangeal [PIP] joints) and by severity of the primary joint contracture (ie, up to 50° or >50° for MP joints and up to 40° or >40° for PIP joints) and then randomized in a 2:1 ratio to either AA4500 0.58 mg or placebo. Upon completion of the double-blind phase (ie, 90-day evaluation after the first injection), all subjects were eligible to enter the open-label extension phase of the study in which they were followed for an additional nine months. Subjects who required further treatment because they either did not achieve reduction in contracture to 5° or less, the cord affecting the primary joint received placebo, another cord received less than three injections of AA4500, or they had untreated cords that were affecting other joints had the option to receive up to five additional injections of AA4500 0.58 mg in the open-label extension phase, with individual cords receiving up to three injections of AA4500.

This study was designed to be part of the larger clinical program, for adult patients with Dupuytren's contracture with a palpable cord, where the data from 2 pivotal Placebo-Controlled studies (AUX-CC-857 [NCT00528606] and AUX-CC-859 [NCT00533273]) and 7 non-pivotal studies were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of advanced Dupuytren's disease, with a fixed flexion deformity of at least one finger, other than the thumb, that had a contracture at least 20°, but not greater than 100°, for MP (80° for PIP) joints, caused by a palpable cord.
* Had a positive "table top test," defined as the inability to simultaneously place the affected finger(s) and palm flat against a table top.
* Were naive to AA4500 treatment
* Were judged to be in good health, based upon the results of a medical history, physical examination, and safety laboratory profile.

Exclusion Criteria:

* Had a chronic muscular, neurological, or neuromuscular disorder that affected the hands.
* Had received a treatment for advanced Dupuytren's disease, including surgery (fasciectomy or surgical fasciotomy), needle aponeurotomy/fasciotomy, or injection of verapamil and/or interferon on the selected primary joint within 90 days before the first dose of study drug.
* Had a known recent history of stroke, bleeding, a disease process that affected the hands, or other medical condition, which in the investigator's opinion, would make the subject unsuitable for enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD, Study Director — Endo Pharmaceuticals
Locations (7):
- Australia (7):
  - Rivercity Research, Auchenflower, Queensland
  - Brisbane Hand & Upper Limb Clinic, Brisbane, Queensland
  - Caboolture Clinical Research Centre, Caboolture, Queensland
  - Peninsula Clinical Research Centre, Kippa-Ring, Queensland
  - Menzies Reserarch Institute, Hobart, Tasmania
  - Emeritus Research, Malvern, Victoria
  - Royal Perth Hospital, Shenton Park, Western Australia

REFERENCES:
- See also: XIAFLEX Prescribing Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2010/125338lbl.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500 0.58 mg: Collagenase clostridium histolyticum 0.58 mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints
- Placebo: Placebo (Sucrose and Tris) injection
Period: Double-blind
Arm/Group | AA4500 0.58 mg | Placebo
Started | 45 | 21
Completed | 45 | 19
Not Completed | 0 | 2
Not completed — Withdrew consent | 0 | 2
Period: Open-label
Arm/Group | AA4500 0.58 mg | Placebo
Started | 64 (open-label was extension of double-blind; 64 of 66 patients continued into open-label) | 0 (no placebo - this phase was open label)
Completed | 58 | 0
Not Completed | 6 | 0
Not completed — Withdrawal by Subject | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- AA4500 0.58 mg: Collagenase clostridium histolyticum 0.58 mg injected into MP and/or PIP joints
- Total: Total of all reporting groups
Arm/Group | AA4500 0.58 mg | Placebo | Total
Number analyzed (Participants) | 45 | 21 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 9 | 34
  >=65 years | 20 | 12 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (7.8) | 65.5 (11.1) | 63.8 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 39 | 17 | 56
Race/Ethnicity, Customized [Number; unit: participants]
  White | 45 | 21 | 66
Region of Enrollment [Number; unit: participants]
  Australia | 45 | 21 | 66

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Primary Joint Contracture to 5° or Less
Description: Successfully treated or clinical success in primary joint defined as reduction in contracture to within 0-5° of normal within 30 days of injection.
Time Frame: Within 30 days after last injection
Population: Subjects who were randomized and received at least 1 injection
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 45 | 21
Number analyzed (Joints) | 45 | 21
Percentage of Joints | 44.4 | 4.8
Statistical Analysis 1: Comparison: AA4500 0.58 mg vs Placebo; Test type: Superiority; p < .001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Clinical Improvement in Primary Joint After the Last Injection
Description: Clinical improvement in primary joint defined as ≥50% reduction from baseline in the degree of contracture within 30 days after injection
Time Frame: Baseline, Within 30 days after last injection
Population: Subjects who were randomized and received at least 1 injection
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 45 | 21
Number analyzed (Joints) | 45 | 21
Percentage of Joints | 77.8 | 14.3
Statistical Analysis 1: Comparison: AA4500 0.58 mg vs Placebo; Test type: Superiority; p < .001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percent Reduction From Baseline Contracture of Primary Joint After the Last Injection
Description: Percent change in degree of contracture of primary joint measured as 100 * (baseline contracture - last available post-injection contracture)/baseline contracture
Time Frame: Baseline, Day 30 after last injection
Population: Subjects who were randomized and received at least 1 injection
Measure: Mean (Standard Deviation); unit: Percentage of change
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 45 | 21
Number analyzed (Joints) | 45 | 21
Percentage of change | 70.5 (29.21) | 13.6 (26.10)
Statistical Analysis 1: Comparison: AA4500 0.58 mg vs Placebo; Test type: Superiority; p < .001, ANOVA

4. Secondary Outcome: Change From Baseline Range of Motion in Primary Joint After the Last Injection
Description: Change in degree of range of motion in primary joint measured as last available post-injection range of motion - baseline range of motion
Time Frame: Baseline, Day 30 after last injection
Population: Subjects who were randomized and received at least 1 injection
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 45 | 21
Number analyzed (Joints) | 45 | 21
Degrees | 35.4 (17.77) | 7.6 (14.88)
Statistical Analysis 1: Comparison: AA4500 0.58 mg vs Placebo; Test type: Superiority; p < .001, ANOVA

5. Secondary Outcome: Time to Reach Clinical Success in Primary Joint
Description: Clinical success in primary joint defined as reduction in contracture to within 0-5° of normal within 30 days of injection, displayed in post injection time point categories
Time Frame: Within 30 days after last injection
Population: Subjects who were randomized and received at least 1 injection
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 45 | 21
Number analyzed (Joints) | 45 | 21
Percentage of Joints
  Injection 1, Day 1 | 2.2 | 0.0
  Injection 1, Day 7 | 6.7 | 4.8
  Injection 1, Day 30 | 17.8 | 0.0
  Injection 2, Day 1 | 0.0 | 0.0
  Injection 2, Day 7 | 4.4 | 0.0
  Injection 2, Day 30 | 8.9 | 0.0
  Injection 3, Day 1 | 4.4 | 0.0
  Injection 3, Day 7 | 0.0 | 0.0
  Injection 3, Day 30 | 0.0 | 0.0
  Did not reach Clinical Success | 55.6 | 95.2

6. Secondary Outcome: Clinical Success in Primary Joint After the First Injection
Description: Clinical success in primary joint defined as reduction in contracture to within 0-5° of normal within 30 days of injection.
Time Frame: Within 30 days after first injection
Population: Subjects who were randomized and received at least 1 injection
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 45 | 21
Number analyzed (Joints) | 45 | 21
Percentage of Joints | 26.7 | 4.8
Statistical Analysis 1: Comparison: AA4500 0.58 mg; Test type: Superiority; p = .014, Cochran-Mantel-Haenszel

7. Secondary Outcome: Clinical Improvement in Primary Joint After the First Injection
Description: as for outcome 2
Time Frame: Baseline, Within 30 days after first injection
Population: Subjects who were randomized and received at least 1 injection
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 45 | 21
Number analyzed (Joints) | 45 | 21
Percentage of Joints | 60.0 | 4.8
Statistical Analysis 1: Comparison: AA4500 0.58 mg vs Placebo; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel

8. Secondary Outcome: Percent Reduction From Baseline Contracture of Primary Joint After the First Injection
Description: Percent change in degree of contracture of primary joint measured as 100 * (baseline contracture - last available post-injection contracture prior to next injection)/baseline contracture
Time Frame: Baseline, Day 30 after first injection
Population: Subjects who were randomized and received at least 1 injection
Measure: Mean (Standard Deviation); unit: Percentage of change
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 45 | 21
Number analyzed (Joints) | 45 | 21
Percentage of change | 58.5 (31.74) | 6.0 (20.79)
Statistical Analysis 1: Comparison: AA4500 0.58 mg vs Placebo; Test type: Superiority; p < .001, ANOVA

9. Secondary Outcome: Change From Baseline Range of Motion in Primary Joint After the First Injection
Description: Change in degree of range of motion in primary joint measured as last available post-injection range of motion prior to the next injection - baseline range of motion
Time Frame: Baseline, Day 30 after first injection
Population: Subjects who were randomized and received at least 1 injection
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 45 | 21
Number analyzed (Joints) | 45 | 21
Degrees | 28.6 (17.41) | 3.6 (9.51)
Statistical Analysis 1: Comparison: AA4500 0.58 mg vs Placebo; Test type: Superiority; p < .001, ANOVA

10. Secondary Outcome: Reduction in Non-primary Joint Contracture to 5° or Less After the Last Injection
Description: Successfully treated or clinical success in non-primary joint defined as reduction in contracture to within 0-5° of normal within 30 days of injection.
Time Frame: Within 30 days after last injection
Population: Includes evaluable non-primary joints treated with AA4500 with baseline fixed flexion contracture >5° and at least 1 post-injection contracture measurement in subjects who received at least 1 non-primary joint injection in either study period
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 63
Number analyzed (Joints) | 89
Percentage of Joints | 53.9

11. Secondary Outcome: Clinical Improvement in Non-Primary Joint After the Last Injection
Description: Clinical improvement in non-primary joint defined as ≥50% reduction from baseline in the degree of contracture within 30 days after injection
Time Frame: Baseline, Within 30 days after last injection
Population: as for outcome 10
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 63
Number analyzed (Joints) | 89
Percentage of Joints | 70.8

12. Secondary Outcome: Percent Reduction From Baseline Contracture of Non-Primary Joint After the Last Injection
Description: Percent change in degree of contracture of non-primary joint measured as 100 * (baseline contracture - last available post-injection contracture)/baseline contracture
Time Frame: Baseline, Day 30 after last injection
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of change
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 63
Number analyzed (Joints) | 89
Percentage of change | 66.4 (34.63)

13. Secondary Outcome: Change From Baseline Range of Motion in Non-Primary Joint After the Last Injection
Description: Change in degree of range of motion in non-primary joint measured as last available post-injection range of motion - baseline range of motion
Time Frame: Baseline, Day 30 after last injection
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 63
Number analyzed (Joints) | 89
Degrees | 25.2 (16.80)

14. Secondary Outcome: Time to Reach Clinical Success in Non-Primary Joint
Description: Clinical success in non-primary joint defined as reduction in contracture to within 0-5° of normal within 30 days of injection, displayed in post injection time point categories
Time Frame: Within 30 days after last injection
Population: as for outcome 10
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 63
Number analyzed (Joints) | 89
Percentage of Joints
  Injection 1, Day 1 | 6.7
  Injection 1, Day 7 | 18.0
  Injection 1, Day 30 | 11.2
  Injection 2, Day 0 | 0.0
  Injection 2, Day 1 | 9.0
  Injection 2, Day 7 | 2.2
  Injection 2, Day 30 | 4.5
  Injection 3, Day 0 | 0.0
  Injection 3, Day 1 | 0.0
  Injection 3, Day 7 | 0.0
  Injection 3, Day 30 | 2.2
  Did not reach Clinical Success | 46.1

15. Secondary Outcome: Clinical Success in Non-Primary Joint After the First Injection
Description: Clinical success in non-primary joint defined as reduction in contracture to within 0-5° of normal within 30 days of injection.
Time Frame: Within 30 days after first injection
Population: as for outcome 10
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 63
Number analyzed (Joints) | 89
Percentage of Joints | 36.0

16. Secondary Outcome: Clinical Improvement in Non-Primary Joint After the First Injection
Description: as for outcome 11
Time Frame: Baseline, Within 30 days after first injection
Population: as for outcome 10
Measure: Number; unit: Percentage of Joints
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 63
Number analyzed (Joints) | 89
Percentage of Joints | 58.4

17. Secondary Outcome: Percent Reduction From Baseline Contracture of Non-Primary Joint After the First Injection
Description: Percent change in degree of contracture of non-primary joint measured as 100 * (baseline contracture - last available post-injection contracture prior to next injection)/baseline contracture
Time Frame: Baseline, Day 30 after first injection
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of change
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 63
Number analyzed (Joints) | 89
Percentage of change | 54.7 (38.37)

18. Secondary Outcome: Change From Baseline Range of Motion in Non-Primary Joint After the First Injection
Description: Change in degree of range of motion in non-primary joint measured as last available post-injection range of motion prior to the next injection - baseline range of motion
Time Frame: Baseline, Day 30 after first injection
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 63
Number analyzed (Joints) | 89
Degrees | 20.5 (17.52)

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (non-SAEs) were collected from time of study drug administration, serious adverse events (SAEs) were collected from time subject signed ICF. Non-SAEs & SAEs were collected until 30 days after completion or discharge from study.
Description: This study was designed to be part of the larger clinical program. For information regarding XIAFLEX-associated Serious and Non-serious Adverse events please refer to the XIAFLEX Medication Guide & XIAFLEX Prescribing Information (see links above)
Groups:
- AA4500 0.58 mg: collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints
- Placebo: Placebo injection is comprised of sucrose and Tris
Arm/Group | AA4500 0.58 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 7/63 | 1/21
Other Adverse Events (participants affected / at risk) | 63/63 | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.58 mg (N=63) | Placebo (N=21)
Abdominal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's contracture operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Inguinal hernia repair (Social circumstances) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Orbital cyst (Eye disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.58 mg (N=63) | Placebo (N=21)
Axillary pain (Musculoskeletal and connective tissue disorders) | 8 (11) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 46 (136) | 2 (4)
Dizziness (Nervous system disorders) | 5 (5) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 2 (3)
Injection site haemorrhage (General disorders) | 27 (76) | 0 (0)
Injection site pain (General disorders) | 28 (61) | 2 (3)
Injection site swelling (General disorders) | 23 (55) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 13 (21) | 0 (0)
Oedema peripheral (General disorders) | 54 (163) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36 (82) | 3 (4)
Paraesthesia (Nervous system disorders) | 5 (6) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (26) | 0 (0)
Tenderness (General disorders) | 20 (24) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (2)
Injection site vesicles (General disorders) | 5 (5) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Auxilium Pharmaceuticals, Inc. agreements may vary with individual investigators but will not prohibit any investigator from publishing. Auxilium supports the publication of results from all centers of a multicenter trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.